CLINICAL TRIAL: NCT06417619
Title: The Effect of Mindfulness-Based Psychoeducation on the Mindfulness, Cognitive Defusion and Depression Level of Depression Patients
Brief Title: The Effect of Mindfulness-Based Psychoeducation
Acronym: Mindfulness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Rabia Arpaci, Principal Investigator, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Depression Patients
Record Dates: First submitted 2024-04-09; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Depressive Disorder, Major
Keywords: Depression; Mindfulness; Cognitive Defusion
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled experimental study (Interventional Study Model)
Who Masked: Participant
Masking Description: Participant (Major depression patients)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Mindfulness-based psychoeducation will be implemented in the experimental group in the form of group sessions once a week for a total of 8 weeks. Post-tests will be administered immediately after the completion of psychoeducation sessions for the experimental group, and a follow-up test will be conducted 3 months after the post-test.
  Interventions: Behavioral: Mindfulness-Based Psychoeducation
- Depression Patients (No Intervention): No intervention will be applied to the control group other than routine treatment. For the control group, no intervention will be made, and post-tests will be administered 8 weeks after the pre-test, followed by a follow-up test 3 months after the post-test.

INTERVENTIONS:
Behavioral: Mindfulness-Based Psychoeducation — The Effect of Mindfulness-Based Psychoeducation on Depression Level of Depression Patients
  Arms: Patients

SUMMARY:
This study is a randomized controlled experimental study conducted to determine the effect of mindfulness-based psychoeducation on levels of mindfulness, cognitive defusion, and depression in patients with depression. The sample of the study will consist of 60 patients (30 experimental, 30 control) diagnosed with major depression, recruited from a state hospital. Mindfulness-based psychoeducation will be applied to the experimental group once a week for a total of 8 weeks in the form of group sessions. No intervention other than routine treatment will be applied to the control group.

The primary questions that the study aims to answer are as follows:

Does mindfulness-based psychoeducation increase levels of mindfulness and cognitive defusion in depression patients? Does mindfulness-based psychoeducation decrease levels of depression in depression patients?

DETAILED DESCRIPTION:
In this research, the sample size calculation was performed using the G Power program by conducting a priori power analysis. Previous studies were reviewed and using the Beck Depression Inventory, expected confidence intervals were determined. With a confidence interval of α=0.05 and a test power (1-β) of 0.95, with an effect size of d=0.9632193, a total of 60 patients were calculated, with 30 patients in the experimental group and 30 patients in the control group. Participants included in the study will be assigned to experimental or control groups using block randomization.

Inclusion Criteria for Participation in the study:

Individuals who are literate.Individuals are willing to participate in the study voluntarily.

Individuals without any communication barriers. Individuals aged between 18 and 65 years. Outpatients being followed up with a diagnosis of major depressive disorder according to DSM-5 criteria. Individuals who have not participated in a mindfulness-based psychoeducation program for their illness in the last 5 years.

Exclusion Criteria for Participation in the study:

Individuals diagnosed with comorbid psychiatric disorders. Patients with intellectual impairment (e.g., intellectual disability) or cognitive conditions that make collaboration impossible, such as dementia.

Patients with psychotic symptoms in addition to the depressive picture. Illiterate individuals. Individuals who do not consent to an interview. Individuals receiving inpatient treatment

ELIGIBILITY:
Inclusion Criteria:

* Those who are literate.
* Those willing to participate in the study voluntarily.
* Those without any communication barriers.
* Those aged between 18 and 65 years.
* Outpatients being followed up with a diagnosis of major depressive disorder according to DSM-5 criteria.
* Those who have not participated in a mindfulness-based psychoeducation program for their illness in the last 5 years.

Exclusion Criteria:

* Those diagnosed with another comorbid mental illness
* Patients with mental conditions that make cooperation impossible, such as intellectual impairment (mental retardation) or dementia
* Patients with psychotic symptoms in addition to depression illiterate people
* Patients who do not consent to the interview
* Those receiving inpatient treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The Personal Information Data Form baseline and 2 months | 2 months
  The Personal Information Data Form prepared by the researcher will consist of a total of 10 questions (gender, age, education level, marital status, employment status, income level, cohabitation status, history of hospitalization, history of suicide attempt, medication use, and adherence to treatment).
Beck Depression Inventory baseline and 2 months | 2 months
  The Beck Depression Inventory, developed by Beck et al. (1961), is designed to measure the risk of depression, level of depressive symptoms, and changes in severity in adults (Beck et al., 1961). The Turkish adaptation of the Beck Depression Inventory was conducted by Hisli (1988). The Beck Depression Scale consists of 21 items, each with four options. Each item scores from 0 to 3. Depression score is obtained by summing these scores. The highest possible score is 63, and a higher total score indicates greater severity of depression. A depression score of 17 or higher indicates depression above normal levels
Mindfulness Scale baseline and 2 months | 2 months
  The Mindfulness Scale was developed by Brown and Ryan (2003) (Brown & Ryan, 2003). The Turkish validity and reliability of the scale were conducted by Özyeşil et al. (2011). The scale was designed to measure the overall level of awareness of skills in daily life and attentiveness to them. The scale consists of 15 items, rated on a six-point Likert scale.The scale is also unifactorial, yielding a single score. The lowest possible score on the scale is 15, and the highest is 90. An increase in the score indicates a higher level of mindfulness awareness in individuals.
Drexel Cognitive Defusion Scale baseline and 2 months | 2 months
  Drexel Cognitive Defusion Scale: The Drexel Cognitive Defusion Scale was developed by Forman et al. (2012) to measure the ability to distance oneself from emotions and thoughts (Forman et al., 2012). The scale consists of 10 items rated on a 6-point Likert scale (0: None; 1: A little, 2: To some extent, 3: Moderate level, 4: Quite a lot, 5: A lot). It is possible to calculate a total score from the scale, where higher scores indicate a higher ability to distance oneself from internal emotions and thoughts.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided